CLINICAL TRIAL: NCT04082806
Title: Memory Enhancement by Gamma-hydroxybutyrate vs. Trazodone in Major Depressive Disorder.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Erich Seifritz (Other)
Responsible Party: Sponsor-Investigator, Erich Seifritz, Head of department for psychiatry, psychotherapy and psychosomatic, Psychiatric University Hospital, Zurich
Organization: Psychiatric University Hospital, Zurich (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: Mem-GHB-TRA-Study
Record Dates: First submitted 2019-08-28; First posted 2019-09-09 (Actual); Last update posted 2022-05-12 (Actual); Status verified 2022-05

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Trazodone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- healthy controls (Experimental)
  Interventions: Drug: GHB; Drug: Trazodone; Drug: Placebos
- Major Depressive Disorder (Experimental)
  Interventions: Drug: GHB; Drug: Trazodone; Drug: Placebos

INTERVENTIONS:
Drug: GHB — 50 mg/kg GHB at one experimental night
Drug: Trazodone — 1.5 mg/kg trazodone at one experimental night
Drug: Placebos — placebo oral solution (placebo for GHB) and placebo pills (placebo for trazodon)

SUMMARY:
30 healthy adults and 30 patients with major depressive disorder, will take part in three single-application pharmacological interventions (GHB vs. Trazodone vs. placebo p.o.) to test potential effects of these drugs on nocturnal memory consolidation. All participants will be assessed with mood state questionnaires, tests of emotional, procedural and declarative memory consolidation, polysomnography, EEG and neuroinflammatory biomarkers. At experimental nights, learning tasks are performed prior to sleep. The next morning, recalling tasks are performed. Each subject will pass through 5 study nights (1 screening, 1 adaptation and 3 experimental nights).

ELIGIBILITY:
Arm 1 (healthy controls):

* Healthy participants,
* Non-smoker,
* Age 20-65 years

Arm 2 (patients with depression):

* Diagnosis of major depression (DSM-V),
* Selective Serotonin-Reuptake-Inhibitor (SSRI) or Selective Serotonin-Noradrenalin-Reuptake-Inhibitor (SSNRI) medication,
* Age 20-65 years

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2020-08-06 (Actual); Primary Completion 2022-04-06 (Actual); Study Completion 2022-04-06 (Actual)

PRIMARY OUTCOMES:
slow wave sleep amount | 1 night
  slow wave sleep time (minutes) during the experimental night
performance in emotional memory consolidation tasks by Emotional Picture Memory Task (EPMT) | 10 hours after encoding
  results in EPMT are measured as number of recognized pictures (1-150)
performance in procedural memory consolidation tasks by Finger Sequence-Tapping Task (FSTT) | 10 hours after encoding
  results in FSTT are measured as number of correct sequences typed in 30seconds
performance in declarative memory consolidation tasks by Paired Word List Task (PAWL) | 10 hours after encoding
  Results in PAWL are expressed as number of correct word pairs recalled (1-40).
Blood levels of Brain Derived Neurotrophic Factor (BDNF). | 9 hours after solid drug administration
  Assessed in serum samples collected by venipuncture using a butterfly needle. Unit of measure as blood concentration (ng/l or mg/ml)
homeostatic sleep pressure by Psychomotor Vigilance Task | 10 hours after solid drug administration
  Results are measured in number of correct answers
homeostatic sleep pressure by N-back Task | 10 hours after solid drug administration
  Results are measured in number of correct answers

SECONDARY OUTCOMES:
Sleep quality assessed by Morgen Questionionnaire (MQ) | at 8:00 a.m. after experimental night 1,2 and 3
  structured interview about sleep quality on the previous night. Subjektive sleep time will be assessed in minutes (0-480 minutes). Long sleep time will be a good outcome. Interview time of 5minutes.
Sleep quality assessed by Karolinska Schläfrigkeitsskala (SKK) | at 8:00 a.m. after experimental night 1,2 and 3
  Subjects will report their subjective sleep pressure in a 1-10 points scale. Low values mean low sleep pressure and better therapy response.
Cortisol Saliva Response (CAR) | 0minutes, 15minutes, 30minutes, 45minutes and 60minutes after awekening
  Cortisol concetration in Saliva (nmol/l)
Score on Positive and Negative Affect Schedule (PANAS) | 8 hours after solid drug administration
  self-report questionnaire that consists of two 10-item scales to measure both positive and negative affect. Each item is rated on a 5-point scale of 1 (not at all) to 5 (very much)

CONTACTS AND LOCATIONS:
Locations (1):
- Psychiatric University Hospital, Zurich, Canton of Zurich, Switzerland